CLINICAL TRIAL: NCT05402722
Title: A Phase II Study of Eribulin in Combination With Anti-PD-1 Antibody in Patients With Metastatic Triple-Negative Breast Cancer
Brief Title: Study of Eribulin in Combination With Anti-PD-1 Antibody in Patients With Metastatic Triple-Negative Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Beijing 302 Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: breast-202204
Record Dates: First submitted 2022-04-13; First posted 2022-06-02 (Actual); Last update posted 2022-06-02 (Actual); Status verified 2022-01

CONDITIONS: TNBC - Triple-Negative Breast Cancer
Keywords: TNBC; Eribulin; anti-PD-1 antibody
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — eribulin; spartalizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Eribulin in combination with anti-PD-1 antibody (Experimental): Participants receive eribulin1.4mg/m2 and anti-PD-1 antibody intravenously (IV) every 3 weeks (Q3W) .
  Interventions: Drug: Eribulin; Drug: anti-PD-1 antibody

INTERVENTIONS:
Drug: Eribulin — Eribulin Mesylate，1.4mg/m2，Intravenous infusion，d1，d8，3-week cycle
  Other Names: Halaven
Drug: anti-PD-1 antibody — Sintilimab Injection，Intravenous infusion，200mg，3-week cycle

SUMMARY:
To evaluate the efficacy of Eribulin in Combination With Anti-PD-1 Antibody in Patients With Metastatic Triple-Negative Breast Cancer.

ELIGIBILITY:
Inclusion Criteria:

1. The patients sign the written informed consent.
2. Women aged 18-75.
3. The pathologic diagnosis of unresectable recurrent or metastatic triple-negative breast cancer ［ER-negative(IHC<1%), PR-negative(IHC<1%), HER2-negative（IHC-/+ or IHC++ and FISH/CISH-）］. Patients with at least one measuring lesion that was conformed to RECIST v1.1 standard.
4. PD-1/PD-L1positive or TMB≥5.
5. Prior therapy (adjuvant/neoadjuvant/advanced) must have included an anthracycline and/or a taxane in any combination or order and either in the early or metastatic disease setting unless contraindicated for a given patient.
6. Eastern Cooperative Oncology Group (ECOG) performance status of ≤ 1.
7. The results of patient's blood tests are as follows:

   • Hb≥90g/L; • Plt≥100^9/L; • Serum albumin ≥3g/dL;• Neutrophils≥1.5^9/L; TSH≤ normal upper limit (ULN);• ALT and AST ≤1.5 ULN (liver metastases ≤3 ULN); • TBIL ≤ULN (total bilirubin ≤1.5 ULN in Gilbert's syndrome or liver metastasis subjects);• ALT and AST ≤1.5 ULN (liver metastases ≤3 ULN);• AKP≤ 2.5 ULN; • Renal function within 7 days before the first administration: serum creatinine ≤1.5 ULN or creatinine clearance ≥60mL/min
8. Female subjects of childbearing potential must have a negative serum pregnancy test within 7 days before the first dose and must be willing to use very efficient barrier methods of contraception for the course of the study through 6 months after the last dose of study treatment.

Exclusion Criteria:

1. The subjects had a central nervous system metastases with clinical symptoms.
2. Subjects with treatment history of PD-1 / PD-L1 inhibitors;
3. Peripheral neuropathy ≥ grade 2; Cardiac dysfunction, hyperthyroidism or hypothyroidism, type 1 diabetes, active hepatitis and tuberculosis; Autoimmune diseases requiring systemic treatment, and a history of pneumonia (requiring corticosteroid treatment) or interstitial lung disease.
4. Pregnant or lactating women.
5. Other clinical trials of drugs were used in the first four weeks before the first dose.
6. The subjects had any history of autoimmune disease or any use of systemic glucocorticoid or immunosuppressive medications.
7. Hereditary or acquired bleeding and thrombotic tendencies (such as hemophilia, coagulation dysfunction, thrombocytopenia, hypersplenism, etc.).
8. Congenital or acquired immune deficiency (such as HIV infection);
9. Receive live vaccine within 4 weeks before or during the study period;
10. Patients who are allergic to or contraindicated to the experimental drugs.
11. Other malignant tumors in the past, except cervical cancer and non melanoma skin cancer, which have survived for 5 years without disease.
12. Subjects with any other diseases that are unfit for the treatment.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 30 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-12-31 (Estimated); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival，PFS | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
  The time from the date of randomization to the date of first documented progression or date of death from any cause, whichever came first.

SECONDARY OUTCOMES:
Number of participants with Adverse Events | From date of treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
  Adverse Events are monitored throughout the trial and for 30 days after discontinuation of treatment (90 days for serious adverse events) and graded according to the Common Terminology Criteria for Adverse Events, version 4.0, of the National Cancer Institute.
the correlation between the expression of PD-L1 of circulating tumor cells and prognosis | From one week before treatment until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 10 months
  To detect the differences of the expression of PD-L1 in patients with different curative effects and prognosis,including the number of circulating tumor cells,and PD-L1 expression or others.

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Medical Center of PLA General Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes